CLINICAL TRIAL: NCT06442111
Title: The Role of Intravenous Ferritin in Optimizing Postoperative Recovery Following Pancreaticoduodenectomy: A Multicenter, Randomized, Controlled Trial
Brief Title: The Role of Intravenous Ferritin in Optimizing Postoperative Recovery Following Pancreaticoduodenectomy
Acronym: Ferritin
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Taeho Hong, Professor, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Seoul_IDA
Record Dates: First submitted 2024-05-12; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Pancreaticojuodenectomy
Keywords: Iron-deficiency anemia; Ferric carboxymaltose; perioperative outcome
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group (Experimental): inclusion criteria : patients with periampullary tumor for whom pancreaticoduodenectomy is planned.
  Interventions: Drug: The intravenous ferritin group; Drug: The placebo group
- The placebo group (Experimental): inclusion criteria : patients with periampullary tumor for whom pancreaticoduodenectomy is planned.
  Interventions: Drug: The intravenous ferritin group; Drug: The placebo group

INTERVENTIONS:
Drug: The intravenous ferritin group — Administer intravenous ferritin approximately 3-7 days before surgery (0.9% normal saline 250ml + 1000 mg of ferric carboxymaltose [Ferinject™, Vifor Pharma, Glattbrugg, Dwitzerland], inject over 15 minutes)
Drug: The placebo group — Administer intravenous 10ml of normal saline (Isotonic Sodium Chloride Injection Daihan(50mL/bag)) approximately 3-7 days before surgery

SUMMARY:
Iron deficiency anemia is well known as a risk factor that worsens postoperative morbidity and patient prognosis. Several studies have shown that intravenous iron administration before surgery is effective in reducing the risk of iron deficiency anemia and improving the postoperative prognosis. However, the risk of iron deficiency anemia after surgery is increased due to the resection of the duodenum, the main organ for iron absorption. Very few studies have been conducted on the postoperative effects of higher pancreatoduodenectomy.

Observe changes in hematological parameters in patients who underwent pancreaticoduodenectomy due to periampullary tumor and confirm the role of intravenous iron supplementation in optimizing postoperative recovery.

DETAILED DESCRIPTION:
Iron deficiency anemia (IDA) has multifactorial causes, including bleeding, insufficient iron absorption, and anemia related to malignant tumors or chronic diseases, which are cytokine-mediated diseases, and is a disease commonly observed in cancer patients. Since cancer surgery generally involves wide resection and tissue manipulation for radical lymph node dissection, systemic inflammation may occur after surgery. This may increase the risk of IDA in patients undergoing surgery by inducing a key regulator of systemic iron hemostasis that impairs intestinal iron absorption.

Pancreaticoduodenectomy, a representative surgery for periampullary neoplastic lesions, is a major surgery accompanied by moderate bleeding and large-scale tissue damage, which predisposes to IDA, and is highly likely to be accompanied by severe bleeding and blood transfusion. The perioperative blood transfusion rate has decreased with the advancement of surgical instruments and techniques, but still remains high at up to 60%. Moreover, since pancreaticoduodenectomy inevitably removes the duodenum, which absorbs iron into the body, the iron absorption function is physiologically impaired, making the patient vulnerable to IDA. Additionally, after pancreaticoduodenectomy, oral intake is often lacking for a relatively long period of time due to complex anastomosis. Therefore, the risk of IDA after pancreaticoduodenectomy may be very high regardless of the presence or absence of preoperative anemia.

IDA is a well-known risk factor for postoperative morbidity and poor prognosis of postoperative patients, and allogeneic transfusion to correct anemia is associated with an increased risk of developing infectious and non-infectious complications, including cancer recurrence, cardiac complications, and prolonged hospitalization. Available.

Research results are currently being published showing that correcting anemia through preoperative intravenous iron injection can improve the patient's postoperative prognosis. In the field of colon or heart surgery, the effect of preventing the occurrence of IDA in people diagnosed with IDA before surgery has been reported. In particular, in patients with postoperative anemia, serum hemoglobin, ferritin, and transferrin saturation levels improved rapidly, and indiscriminate blood transfusion was prevented. Another study showed that it was effective in reducing postoperative blood transfusion and intensive care unit length of stay in elderly patients. However, there is a lack of research on the effect of preoperative iron injections on postoperative clinical outcomes after pancreatoduodenectomy, where most patients are elderly and have high intraoperative bleeding.

Therefore, the purpose of this study was to evaluate changes in hematological parameters in patients who underwent pancreaticoduodenectomy due to periampullary lesions and their effect on improving clinical outcomes within 12 weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients who diagnosed periampullary tumor
* age under 75, over 18 years

Exclusion Criteria:

1. palliative or emergency surgery,
2. incurable or metastatic disease state,
3. insufficient data,
4. accompanying hematologic disorders that may cause anemia,
5. loss to follow-up,
6. ferritin Contraindications to intravenous administration (pregnancy or lactation, age under 18 years, history of severe asthma or infection, chronic renal failure, simultaneous oral and intravenous iron administration, allergic reaction to iron)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of hemoglobin responders by 12 weeks after surgery | 12 weeks
  If your hemoglobin level increases from baseline to week 12 by more than 2 g/dL or 14 and your hemoglobin level is more than 11 g/dL

SECONDARY OUTCOMES:
Postoperative transfusion rate | 12 weeks
  Postoperative transfusion rate (%) : If blood transfusion is required within 72 hours after surgery
morbidity | 12 weeks
  morbidity (%) : postoperative complications (infectious, non-infectious complications)

CONTACTS AND LOCATIONS:
Overall Officials: Sung eun Park, Study Director — Catholic University Seoul St. Mary's Hospital

IPD SHARING:
Plan to Share IPD: No